CLINICAL TRIAL: NCT00380861
Title: Does Implant Design Improve Postoperative Flexion?A Prospective, Randomized, Comparative, Multi-center Study Comparing PFC® Sigma™ RP Knee Versus PFC® Sigma™ RP-F Implanted in Simultaneous Bilateral Subjects
Brief Title: Does Implant Design Improve Postoperative Flexion?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04092
Record Dates: First submitted 2006-09-26; First posted 2006-09-27 (Estimated); Results first posted 2011-04-05 (Estimated); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Non-inflammatory Arthritis
Keywords: Total Knee Replacement; Flexion; Range of Motion; Activities of Daily Living; Implant design; Subject Satisfaction; Non-inflammatory arthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PFC Sigma RP-F (Active Comparator): PFC® Sigma™ RP-F knee implant is a posterior stabilized cemented component cemented that is implanted with a standard posterior stabilized surgical technique.
  Interventions: Device: Total knee replacement using the PFC Sigma RPF knee implant.
- PFC Sigma RP (Active Comparator): P.F.C.® Sigma™ Rotating Platform (RP) Cruciate Retaining Knee System has a special insert that helps the knee move more like it did before the knee replacement.
  Interventions: Device: Total knee replacement using the PFC Sigma RP knee implant

INTERVENTIONS:
Device: Total knee replacement using the PFC Sigma RPF knee implant. — Total knee replacement
  Arms: PFC Sigma RP-F
Device: Total knee replacement using the PFC Sigma RP knee implant — Total knee replacement
  Arms: PFC Sigma RP

SUMMARY:
This study will evaluate whether design features of one implant design allows more knee bend than the other. Patients will have 1 design in the left knee and 1 design in their right knee. Both knee surgeries will be on the same day.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether the passive, non-weight-bearing flexion is superior with the posterior-stabilized PFC® Sigma™ RP-F compared to the posterior-stabilized PFC® Sigma™ RP in bilateral Subjects receiving both implants and if this difference is a function of implant design.

ELIGIBILITY:
Inclusion Criteria:

* Non-Inflammatory Arthritis
* Age = 40-70 years
* Male or female
* Suitable for devices in study
* Needing primary simultaneous bilateral knee replacements
* Willing to consent and authorize release of personal health information
* Subjects who are able to understand this clinical investigation, co-operate with investigational procedures and are willing to return to the clinic, hospital and predefined physical therapy centers for all the required postoperative follow-ups,

Exclusion Criteria:

* Existing conditions that would compromise participation
* Multiple joint involvement
* Pregnant/lactating women
* Inflammatory arthritis
* Fixed flexion contracture greater than 20 degrees
* Previous knee replacement of any type
* Needing device(s) not specified in protocol
* The Subject is a known drug or alcohol abuser or has a psychological disorder that would compromise follow-up
* Those who have participated in an investigation in the last 3 months
* Those involved in personal injury litigation, medical-legal or workers compensation claims
* Failure to follow surgical technique details specified in the protocol

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2006-03-01 (Actual); Primary Completion 2009-12-01 (Actual); Study Completion 2009-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tammy O'Dell, EMT, CCRA, CCRC, Study Director — DePuy Orthopaedics
Locations (4):
- United States (4):
  - Doug Dennis, Denver, Colorado
  - Heekin Orthopaedics, Jacksonville, Florida
  - University of Iowa Hospital & Clinic Dept. of Orthopaedic Surgery, Iowa City, Iowa
  - Lakewood Orthopaedic Surgeons, Lakewood, Washington

REFERENCES:
- [Derived] Tippett SR, Mang J, Dwyer KA, Lesko J, O'Dell T. Collecting data with Palm technology: comparing preoperative expectations and postoperative satisfaction in patients undergoing total knee arthroplasty. J Bone Joint Surg Am. 2010 Dec;92 Suppl 2:59-67. doi: 10.2106/JBJS.J.00827. No abstract available. PMID 21123592

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were eight clinical investigators participating in the investigation. Subjects who were to receive simultaneous bilateral knee replacement were recruited for this study, where one knee was to receive the PFC Sigma Rotating Platform high flexion (RP-F) device and the other knee was to receive the PFC Sigma Rotating Platform (RP) device. 93 Subjects were enrolled in the study.
Pre-assignment Details: The randomization was a two stage scheme in order to minimize bias that could potentially be introduced due to differences in preoperative range of motion (ROM) between a subject's right and left legs.
Units Other Than Participants: knees
Groups:
- PFC® Sigma™ RP-F, Posterior Stabilized Total Knee Replacement: Comparison of PFC Sigma RP-F design in the one knee to the PFC Sigma RP design in the other knee.
- PFC® Sigma™ RP, Posterior Stabilized Total Knee Replacement: Comparison of PFC Sigma RP design in the one knee to the PFC Sigma RP-F design in the other knee.
Period: Overall Study
Arm/Group | PFC® Sigma™ RP-F, Posterior Stabilized Total Knee Replacement | PFC® Sigma™ RP, Posterior Stabilized Total Knee Replacement
Started | 93; 93 knees | 91; 91 knees (Two subjects received the PFC Sigma RP-F device but not the RP and their results are not included.)
Completed | 75; 75 knees | 74; 74 knees
Not Completed | 18; 18 knees | 17; 17 knees

BASELINE CHARACTERISTICS:
Units Other Than Participants: knees
Groups:
- Total: Total of all reporting groups
Arm/Group | PFC® Sigma™ RP-F, Posterior Stabilized Total Knee Replacement | PFC® Sigma™ RP, Posterior Stabilized Total Knee Replacement | Total
Number analyzed (Participants) | 93 | 91 | 93
Number analyzed (knees) | 93 | 91 | 184
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Subjects have a Sigma RP in one knee and a Sigma RP-F in their other knee
  years | 61.4 (5.6) | 61.4 (5.7) | 61.4 (5.8)
Sex: Female, Male [Count of Units; unit: knees] — Population: there were 61 females and 32 males in the study. Each participant had a Sigma RP in one knee and a Sigma RP-F in the other
  knees
    Female | 61 | 60 | 121
    Male | 32 | 31 | 63
Region of Enrollment [Count of Units; unit: knees]
  United States: United States | 93 | 91 | 184

OUTCOME MEASURES:

1. Secondary Outcome: Subgroup Analysis - Passive Flexion Analyzed and Reported for Pre-op, 6- and 12-months, for Subjects With Less Than 120 Degrees Passive Flexion Pre-op in Either Knee
Description: The patient lies supine (on their back) on the table and a medically trained professional moves the limb to bend the knee to a maximum flexion position. The angle of flexion is measured with a goniometer, which is an angle-measuring device.
Time Frame: Collected at Pre-operative, 2 and 6 weeks and 6- and 12-months, analyzed and reported for pre-op, 6- and 12-months
Measure: Mean (Standard Deviation); unit: Degrees of passive flexion
Units Other Than Participants: Knees
Groups:
- Passive Flexion for Standard Knee Device at Pre-op: Single leg passive flexion for Standard Knee Device at pre-op
- Passive Flexion for Standard Knee Device at 6-months: Single leg passive flexion for Standard Knee Device at 6-months
- Passive Flexion for Standard Knee Device at 12-months: Single leg passive flexion for Standard Knee Device at 12-months
- Passive Flexion for High Flexion Knee Device at Pre-op: Single leg passive flexion High Flexion Knee Device at pre-op
- Passive Flexion for High Flexion Knee Device at 6-months: Single leg passive flexion for High Flexion Knee Device at 6-months
- Passive Flexion for High Flexion Knee Device at 12-months: Single leg passive flexion for High Flexion Knee Device at 12-months
Arm/Group | Passive Flexion for Standard Knee Device at Pre-op | Passive Flexion for Standard Knee Device at 6-months | Passive Flexion for Standard Knee Device at 12-months | Passive Flexion for High Flexion Knee Device at Pre-op | Passive Flexion for High Flexion Knee Device at 6-months | Passive Flexion for High Flexion Knee Device at 12-months
Number analyzed (Participants) | 19 | 16 | 18 | 20 | 17 | 18
Number analyzed (Knees) | 19 | 16 | 18 | 20 | 17 | 18
Degrees of passive flexion | 111.6 (6.0) | 118.9 (13.9) | 120.2 (11.3) | 111.4 (5.8) | 120.9 (12.7) | 124.7 (9.8)

2. Secondary Outcome: Patient Specific Anthropometrics
Description: Various Patient specific anthropometrics were examined to assess their potential influence and interaction on post-op outcomes.
Time Frame: Collected at pre-op
Measure: Mean (Standard Deviation); unit: Centimeters
Groups:
- Thigh Circumference in Centimeters (cm): Thigh circumference was measured 10 cm proximal to the superior aspect of the patella bone
- Ankle Circumference in Centimeters (cm): Ankle circumference was measured in centimeters
- Skin-fold in Centimeters (cm): Skin-fold was measured in the middle of the thigh, 10 cm proximal to the superior patellar pole, using calipers.
Arm/Group | Thigh Circumference in Centimeters (cm) | Ankle Circumference in Centimeters (cm) | Skin-fold in Centimeters (cm)
Number analyzed (Participants) | 93 | 93 | 93
Centimeters | 50.2 (6.3) | 24.8 (2.7) | 3.23 (1.46)

3. Secondary Outcome: American Knee Society (AKS) Score
Description: AKS Score post-op at 12-months is reported for the final visit AKS score is a 0 -100-point scale with 100 being best knee condition.
Time Frame: Collected Pre-operative, 2 and 6 weeks and 6 and 12 months follow up. Reporting for final 12-month interval
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: Knees
Groups:
- AKS for the Standard Knee Device: AKS for the Standard Knee Device at 12-months
- AKS for the High Flexion Knee Device: AKS for the High Flexion Knee Device at 12 months
Arm/Group | AKS for the Standard Knee Device | AKS for the High Flexion Knee Device
Number analyzed (Participants) | 80 | 81
Number analyzed (Knees) | 80 | 81
Units on a scale | 85.6 (11.5) | 87.0 (10.7)

4. Secondary Outcome: KOOS Pain Sub-score
Description: KOOS is a self-reported outcome measure assessing the patient's opinion about health, symptoms, and functionality of their knee. There are 5 sub-scales: symptoms, pain activity of daily living, sports/recreation and quality of life. Further, the sub-score for pain is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems.
Time Frame: Pre-operative, 2 and 6 weeks and 6 and 12 months and analyzed and reported for pre-op, 6- and 12-months follow up
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: Knees
Groups:
- KOOS Pain Sub-score Standard Knee Device at Pre-op: KOOS Pain Sub-score for Standard Knee Device at pre-op. The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems.
- KOOS Pain Sub-score Standard Knee Device at 6-months: KOOS Pain Sub-score for Standard Knee Device at 6-months. The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems.
- KOOS Pain Sub-score Standard Knee Device at 12-months: KOOS Pain Sub-score Standard Knee Device at 12-months. The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems.
- KOOS Pain Sub-score High Flexion Knee Device at Pre-op: KOOS Pain Sub-score High Flexion Knee Device at pre-op. The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems
- KOOS Pain Sub-score High Flexion Knee Device at 6-months: KOOS Pain Sub-score High Flexion Device at 6-months. The score is a percentage score from 0 to 100 with 0 representing extreme problems and 100 representing no problems.
- KOOS Pain Sub-score High Flexion Knee Device at 12-months: KOOS Pain Sub-score High Flexion Knee Device at 12-months. The score is a percentage score from 0 to 100 with 0 representing extreme problems and 100 representing no problems.
Arm/Group | KOOS Pain Sub-score Standard Knee Device at Pre-op | KOOS Pain Sub-score Standard Knee Device at 6-months | KOOS Pain Sub-score Standard Knee Device at 12-months | KOOS Pain Sub-score High Flexion Knee Device at Pre-op | KOOS Pain Sub-score High Flexion Knee Device at 6-months | KOOS Pain Sub-score High Flexion Knee Device at 12-months
Number analyzed (Participants) | 86 | 67 | 79 | 88 | 68 | 80
Number analyzed (Knees) | 86 | 67 | 79 | 88 | 68 | 80
Units on a scale | 45.7 (19.2) | 84.0 (14.8) | 89.5 (14.0) | 45.3 (18.2) | 83.1 (14.9) | 90.0 (11.8)

5. Secondary Outcome: Ability to Perform Activities of Daily Living (ADLs) as Per the KOOS Sub-scale for ADLs
Description: KOOS is a self-reported outcome measure assessing the patient's opinion about health, symptoms, and functionality of their knee. There are 5 sub-scales: symptoms, pain, activity of daily living, sports/recreation and quality of life. The score is a percentage score from 0 to 100 with 0 representing extreme problems and 100 representing no problems.
Time Frame: Collected at pre-operative, 2 and 6 weeks and 6 and 12 months, analyzed and reported for pre-op, 6 and 12-months
Measure: Mean (Standard Deviation); unit: Points on a scale
Units Other Than Participants: Knees
Groups:
- KOOS Sub-scale for Activity of Daily Living (ADL) for Standard Knee Device at Pre-op: KOOS Sub-scale for Activity of Daily Living for Standard Knee Device at pre-op. Scoring range is 0 (worst) to 100 (best)
- KOOS Sub-scale for Activity of Daily Living for Standard Knee Device at 6-months.: KOOS Sub-scale for Activity of Daily Living for Standard Knee Device at 6-months. Scoring range is 0 (worst) to 100 (best)
- KOOS Sub-scale for Activity of Daily Living for Standard Knee Device at 12-months.: KOOS Sub-scale for Activity of Daily Living for Standard Knee Device at 12-months. Scoring range is 0 (worst) to 100 (best)
- KOOS Sub-scale for Activity of Daily Living for High Flexion Knee Device at Pre-op: KOOS Sub-scale for Activity of Daily Living for High Flexion Knee Device at pre-op. Score range is 0 (worst) to 100 (best)
- KOOS Sub-scale for Activity of Daily Living for High Flexion Knee Device at 6-months: KOOS Sub-scale for Activity of Daily Living for High Flexion Knee Device at 6-monhts. Score range is 0 (worst) to 100 (best).
- KOOS Sub-scale for Activity of Daily Living for High Flexion Knee Device at 12-months: KOOS Sub-scale for Activity of Daily Living for High Flexion Knee Device at 12-months. Score range is 0 (worst) to 100 (best).
Arm/Group | KOOS Sub-scale for Activity of Daily Living (ADL) for Standard Knee Device at Pre-op | KOOS Sub-scale for Activity of Daily Living for Standard Knee Device at 6-months. | KOOS Sub-scale for Activity of Daily Living for Standard Knee Device at 12-months. | KOOS Sub-scale for Activity of Daily Living for High Flexion Knee Device at Pre-op | KOOS Sub-scale for Activity of Daily Living for High Flexion Knee Device at 6-months | KOOS Sub-scale for Activity of Daily Living for High Flexion Knee Device at 12-months
Number analyzed (Participants) | 79 | 69 | 75 | 83 | 69 | 75
Number analyzed (Knees) | 79 | 69 | 75 | 83 | 69 | 75
Points on a scale | 49.0 (20.2) | 85.4 (14.0) | 90.4 (11.8) | 47.9 (19.2) | 85.6 (12.7) | 90.1 (11.3)

6. Secondary Outcome: Patellar Crepitus Defined as No Crepitus, FINE or COARSE
Description: Patellar Crepitus (grinding in the knee) analyzed and reported for pre-op, 6-months and 12-months and classified as No Crepitus, FINE or COARSE.
Time Frame: Collected at Pre-operative, 6 weeks and 6 and 12 months
Population: Patellar crepitus is measured by touch with the clinician placing a hand over the knee cap and moving the lower leg from flexion to extension. It is classified as coarse, fine or no crepitus.
Measure: Count of Units; unit: Knees
Units Other Than Participants: Knees
Arm/Group | Patellar Crepitus in Standard (RP) Flexion Cohort at Pre-Op | Patellar Crepitus in High Flexion Cohort (RPF) at Pre-op | Patellar Crepitus in Standard Flexion (RP) Cohort at 6-months | Patellar Crepitus in High Flexion (RPF) Cohort at 6 Months | Patellar Crepitus in Standard Flexion (RP) Cohort at 12-months | Patellar Crepitus in High Flexion (RPF) Cohort at 12-months
Number analyzed (Participants) | 91 | 92 | 74 | 75 | 78 | 78
Number analyzed (Knees) | 91 | 92 | 74 | 75 | 78 | 78
Knees
  NO Crepitus | 15 | 13 | 44 | 41 | 52 | 52
  FINE Crepitus | 31 | 37 | 21 | 29 | 22 | 22
  COARSE Crepitus | 45 | 42 | 9 | 5 | 4 | 4

7. Secondary Outcome: Subject Satisfaction
Description: Secondary objective to compare the pre-op goals and post-op satisfaction through the interpretation of data collected with the use of Palm technology for bilateral knee patients
Time Frame: Collected pre-and post-op, reported at 12-months
Measure: Count of Participants; unit: Participants
Groups:
- All Bilateral Patients Reporting Satisfaction at 12-months After Knee Replacement: All bilateral knee replacement patients participating in the Palm technology to assess satisfaction from pre-op goals to 12-months
Arm/Group | All Bilateral Patients Reporting Satisfaction at 12-months After Knee Replacement
Number analyzed (Participants) | 91
Participants | 84

8. Primary Outcome: Knee Society Passive Flexion at 6 Months
Description: as for outcome 1
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Degrees of passive flexion
Units Other Than Participants: Knees
Arm/Group | PFC® Sigma™ RP-F, Posterior Stabilized Total Knee Replacement | PFC® Sigma™ RP, Posterior Stabilized Total Knee Replacement
Number analyzed (Participants) | 93 | 91
Number analyzed (Knees) | 93 | 91
Degrees of passive flexion | 124.2 (11.2) | 124.0 (10.6)

9. Secondary Outcome: Single Leg Active Flexion (SLAF)
Description: Weight-bearing single leg active flexion (SLAF). A medically trained professional conducts this test using a goniometer, which is an angle-measuring device. Of note, pre-op patients have a lower number because they were unable or unwilling to participate in SLAF due to pain.
Time Frame: Pre-op, 6- and 12-months
Measure: Mean (Standard Deviation); unit: Degrees of flexion
Units Other Than Participants: knees
Groups:
- Single Leg Active Flexsion (SLAF) for the Standard Knee Device at Pre-op: Weight bearing Single Leg Active Flexion (SLAF) for the Standard Knee Device at pre-op
- Single Leg Active Flexion (SLAF) for Standard Knee Device at 6-months: Weight bearing Single Leg Active Flexion (SLAF) for Standard Knee Device at 6-months
- Single Leg Active Flexion (SLAF) for Standard Knee Device at 12-months: Weight bearing Single Leg Active Flexion (SLAF) for Standard Knee Device at 12-months
- Single Leg Active Flexion (SLAF) High Flexion Knee Device at Pre-op: Weight bearing Single Leg Active Flexion (SLAF) for High Flexion Knee Device at pre-op
- Single Leg Active Flexion (SLAF) for the High Flexion Knee Device at 6-months: Weight bearing Single Leg Active Flexion (SLAF) for High Flexion Knee Device at 6-months
- Single Leg Active Flexion (SLAF) for the High Flexion Knee Device at 12-months: Weight bearing Single Leg Active Flexion (SLAF) for the High Flexion Knee Device at 12-months
Arm/Group | Single Leg Active Flexsion (SLAF) for the Standard Knee Device at Pre-op | Single Leg Active Flexion (SLAF) for Standard Knee Device at 6-months | Single Leg Active Flexion (SLAF) for Standard Knee Device at 12-months | Single Leg Active Flexion (SLAF) High Flexion Knee Device at Pre-op | Single Leg Active Flexion (SLAF) for the High Flexion Knee Device at 6-months | Single Leg Active Flexion (SLAF) for the High Flexion Knee Device at 12-months
Number analyzed (Participants) | 27 | 70 | 73 | 31 | 72 | 74
Number analyzed (knees) | 27 | 70 | 73 | 31 | 72 | 74
Degrees of flexion | 124.6 (11.1) | 126.0 (11.0) | 126.6 (10.6) | 120.9 (13.3) | 125.2 (10.8) | 127.5 (11.1)

ADVERSE EVENTS:
Arm/Group | PFC® Sigma™ RP-F, Posterior Stabilized Total Knee Replacement | PFC® Sigma™ RP, Posterior Stabilized Total Knee Replacement
Serious Adverse Events (participants affected / at risk) | 3/93 | 2/91
Other Adverse Events (participants affected / at risk) | 10/93 | 8/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PFC® Sigma™ RP-F, Posterior Stabilized Total Knee Replacement (N=93) | PFC® Sigma™ RP, Posterior Stabilized Total Knee Replacement (N=91)
Infection (Infections and infestations) | 1 (2) | 1 (1)
Loosening (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Polyethylene Failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PFC® Sigma™ RP-F, Posterior Stabilized Total Knee Replacement (N=93) | PFC® Sigma™ RP, Posterior Stabilized Total Knee Replacement (N=91)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 5 (6) | 4 (4)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 8 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less